CLINICAL TRIAL: NCT06854952
Title: A Phase 2 Study to Evaluate the Efficacy, Safety, and Tolerability of TERN-601 in Adults With Overweight or Obesity
Brief Title: A Clinical Study to Evaluate the Efficacy, Safety, and Tolerability of TERN-601 in Adults With Overweight or Obesity
Acronym: FALCON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Terns, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TERN601-2003
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Overweight or Obesity
Keywords: overweight; obesity; obese; glucagon-like peptide-1 receptor agonist; GLP-1 receptor agonist; GLP-1
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TERN-601 Dose 1 (Experimental): Orally administered once daily.
  Interventions: Drug: TERN-601
- TERN-601 Dose 2 (Experimental): Orally administered once daily.
  Interventions: Drug: TERN-601
- TERN-601 Dose 3 (Experimental): Orally administered once daily.
  Interventions: Drug: TERN-601
- TERN-601 Dose 4 (Experimental): Orally administered once daily.
  Interventions: Drug: TERN-601
- Matching Placebo (Placebo Comparator): Orally administered once daily.
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: TERN-601 — Investigational drug
  Arms: TERN-601 Dose 1; TERN-601 Dose 2; TERN-601 Dose 3; TERN-601 Dose 4
Other: Matching Placebo — Matching placebo
  Arms: Matching Placebo

SUMMARY:
This is a Phase 2a multicenter, randomized, double-blind, placebo-controlled clinical trial studying the efficacy, safety, and tolerability of orally administered TERN-601 in adults with overweight or obesity.

ELIGIBILITY:
Key Inclusion Criteria:

1. Female or male aged 18 to 75 years
2. Body mass index (BMI) of:

   1. ≥ 30 kg/m^2 to < 50 kg/m^2

      OR
   2. ≥ 27 kg/m^2 to < 30 kg/m^2 with at least 1 weight-related comorbidity
3. HbA1c < 6.5%
4. Stable self-reported body weight for at least 3 months prior to study (< 5% body weight gain or loss)

Key Exclusion Criteria:

1. Have diabetes mellitus
2. Have obesity induced by medication or other diagnosed endocrinologic disorders
3. Have had or are planning surgical treatment or device-based therapy for obesity
4. Lifetime history of suicide attempt

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Percent Change in Body Weight | 12 weeks
  Percent change (%) in body weight from baseline to Week 12

SECONDARY OUTCOMES:
Change in Body Weight | 12 weeks
  Change in body weight (kg) from baseline to Week 12
≥ 5% Weight Loss | 12 weeks
  Proportion of participants achieving ≥ 5% weight loss

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - FALCON Research Site, Birmingham, Alabama
  - FALCON Research Site, Homewood, Alabama
  - FALCON Research Site, Tucson, Arizona
  - FALCON Research Site, Spring Valley, California
  - FALCON Research Site, Port Orange, Florida
  - FALCON Research Site, Louisville, Kentucky
  - FALCON Research Site, Marrero, Louisiana
  - FALCON Research Site, Boston, Massachusetts
  - FALCON Research Site, Rochester, Minnesota
  - FALCON Research Site, City of Saint Peters, Missouri
  - FALCON Research Site, Beachwood, Ohio
  - FALCON Research Site, Medford, Oregon
  - FALCON Research Site, Dallas, Texas
  - FALCON Research Site, Houston, Texas
  - FALCON Research Site, San Antonio, Texas
  - FALCON Research Site, St. George, Utah
  - FALCON Research Site, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: No